CLINICAL TRIAL: NCT03247933
Title: "Clinical Trial Randomized, Controlled, Parallel-group and Open About the Use of"TELEMEDICINE"in the Management of the Maintenance of a Respiratory Rehabilitation Program Phase in Patients With Chronic Respiratory Diseases"
Brief Title: TELEMEDICINE,Maintenance of a Respiratory Rehabilitation Program in Patients With Chronic Obstructive Pulmonary Disease.
Acronym: TELEREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JUAN B GALDIZ ITURRI (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital de Cruces (Other)
Responsible Party: Sponsor-Investigator, JUAN B GALDIZ ITURRI, PhD- Neumologist, Hospital de Cruces
Organization: Hospital de Cruces (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELEREHAB
Record Dates: First submitted 2015-09-15; First posted 2017-08-14 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: COPD
Keywords: COPD; RESPIRATORY REHABILITATION TELEMEDICINE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Coded databases
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (TeleRR) (Experimental): The intervention: Telemedicine: Maintenance Respiratory Rehabilitation. Patients will receive a personal program of maintenance Respiratory Rehabilitation supported by telemedicine (TeleRR).
  A personal program of Respiratory rehabilitation consists on: 20-30 minutes of static bicycle exercises + 3 series of ten repetitions from 4 different types of exercises with weights / cufflinks. 3 days a week, every week for a year.
  The exercises dates must be sent after doing the training each day by the PDA . The dates will be monitoring by the physician .
  Interventions: Device: Telemedicine: Maintenance Respiratory Rehabilitation
- Clinical Practice (Recommendation) (No Intervention): No intervention. A recommendation from standard maintenance respiratory rehabilitation program with a minimum monitoring.
  Clinical practice.

INTERVENTIONS:
Device: Telemedicine: Maintenance Respiratory Rehabilitation — Telemedicine: Maintenance Respiratory Rehabilitation. Patients will receive a personal program of maintenance respiratory rehabilitation supported by telemedicine (TeleRR).
  A personal program of Respiratory rehabilitation consists on: 20-30 minutes of static bicycle exercises + 3 series of ten repetitions from 4 different types of exercises with weights / cufflinks. 3 days a week, every week for a year.
  They will be in their homes doing the program of treatment prescribed by the physician. They will be provided with the material that is needed: 1 static bicycle, 2-weights / cufflinks, 3-device mobile (smartphone/PDA) + Pulse Oximeter.
  The patient must send the exercises every day that are scheduled training exercises once have been completed.
  Arms: Telemedicine (TeleRR)

SUMMARY:
Respiratory rehabilitation (RR) has been shown to provide benefits in patients with Chronic Obstructive Pulmonary Disease (COPD) with a degree of evidence A.

These benefits are primarily focused on an increase in the capacity of effort for activities of daily living and in an improvement in the quality of life related to health (HRQOL) a constant to the RR critique is the fact that the benefits achieved with programmes are lost in a progressive and constant way once the patient completes the treatment and lost contact with the team.

The introduction of new technologies in different fields of medicine has been a new approach when it comes to the management of various diseases and treatments in chronic patients. In the case of the RR telemedicine provides a new tool.

COPD disease very prevalent and chronic it is generator of a high economic cost. The possibility of universalizing the rehabilitation treatment would involve a potential savings in this population group ,another potential benefit is as translational trial as part of the development of a new technology and its possible application to clinical practice.

General objective: to determine whether a program of TeleRehabilitation (TeleRR)- Respiratory Rehabilitation Maintenance (RRm) after an intensive initial program of RR, is a useful intervention against the current usual strategy (intensive program of RR and a recommendation of not protected maintenance program).

Method: clinical trial , open, randomized, multicenter, parallel group, and focus of superiority with a strategy of Telerehabilitation program respiratory of maintenance after an intensive RR for 8 weeks in patients diagnosed with grade moderately - severe stable COPD (Bode 3-7).

DETAILED DESCRIPTION:
1. SELECTION AND WITHDRAWAL OF SUBJECTS

   1.1 INCLUSION CRITERIA

   To be eligible to participate in this study, subjects must meet the following inclusion criteria:

   Patients diagnosed with COPD aged less than 75 years BODE index of 3-7 clinical stability, understood as not having an exacerbation (*) of the COPD and not require treatment with antibiotics, corticoids systemic and/or hospitalization, at least 1 month prior to inclusion in the study. You have been reported to the subject and has been given sufficient time and opportunity to consider their participation has given its consent in writing. Able to use technology the subject is willing and is able to meet all the requirements of the study.

   (*) Exacerbation: Exacerbation means worsening of two or more of the following main symptoms for at least 2 consecutive days:

   Increase in volume of sputum, sputum Purulence ,Dyspnea

   or

   • Worsening of any main symptom along with one of the following symptoms for at least 2 consecutive days.
   * Resfriado (rinorrea y/o congestión nasal)
   * Fever without any other cause
   * Cough
   * Wheezing

   1.2 Exclusion criteria

   Patients who have any of the following exclusion criteria may not be included in the trial:

   • Presence of osteo-muscular pathology that limit or preclude the exercises. Presence of heart disease which hinders exercise. Patients with bronchiectasis or other respiratory disorders other than COPD. Comorbidity who hinders or blocks the making of respiratory rehabilitation of maintenance program. Less than 2 years life expectancy.

   Any unstable medical or psychiatric process or substance abuse which, in the opinion of the investigator, would affect the ability of the patient to complete the study or impede their participation in the same

   Withdrawal of subjects and procedures criteria

   Patients may leave the study at any time. Each month the researcher will check filling in each patient assigned to the experimental group respiratory rehabilitation program. If a patient does not fill this program for 2 consecutive months, excluding impossibility for clinical situation and medical criteria, will be removed from the study.

   In addition respiratory rehabilitation maintenance in both treatment groups will be suspended if any adverse events that justify it at the discretion of the investigator.

   If so, the follow-up of the patients will continue also to analyze the results according to an intention of treatment strategy.La retirada de los sujetos así como sus motivos quedará reflejada tanto en el historial clínico como en el cuaderno de recogida de datos.

   Any death that occurs during the performance of the EC must be notified immediately to the promoter and the competent Ethics Committee.

   Withdrawals of subjects is not replaced
2. PROTOCOL TREATMENT

The information sheet will be delivered to the patient all of those potentially eligible patients according to the inclusion criteria marked and no exclusion criteria (point 6) let them the time needed to read the document and make all ask them as necessary. If the patient decides to participate in the trial, it will ask you to sign the informed consent form.

SELECTION VISIT

This visit will include the test data for patients diagnosed with COPD, which includes: "history: on the scale of MRC Dyspnoea score" "physical examination: weight, height, body mass index, brachial perimeter crease triceps and quadriceps strength " X-ray of thorax and electrocardiogram respiratory function tests (spirometry, Lung volumes, transfer to CO, maximum respiratory pressure and blood gas capacity) maximum questionnaire of quality of life-related lower-limb exercise test with the Health: CRQ (self-administered version), and SF-36 test of 6 minutes 6 minutes walking test with assessment of breathlessness to the effort using the Borg scale at the beginning and at the end of six minutes the BODE index calculation test

Criteria of Inclusion / Exclusion criteria, information to the patient and informed consent signature, indicating date

On this visit the code of patient will be assigned to each of the patients who accept to participate in the trial and that sign the informed consent

INTENSIVE REHABILITATION (RRi) (8 weeks- ± 4 days)

Once signed the informed consent (CI) the patient will receive an initial program of intensive RR (hospital-based program standard according to usual practice) participate in this phase all the patients in the study and will receive equal treatment. This program will be taught in groups of 5 patients (approx) and will last a total of 8 weeks. Patients will have to go to the hospital 3 hours/d 3 days per week where respiratory rehabilitation program will be intensive.

The program will include the following sections.

1. Education: 4 sessions on knowledge of the disease and medication management learning.
2. General physiotherapy: teach to make the diaphragmatic breathing, drainage of secretions (if applicable) and relaxation techniques.
3. Muscle training:

3.a.-upper extremity muscles: will be weight-bearing exercises. The initial charge will be 500gr and will increase progressively depending on the tolerance of the patient. The training time will be 30 minutes.

3.b.-lower extremity muscles: will be made with an antispasm. The initial charge will be 50% of the maximum load in the progressive stress test. The workload according to the tolerance of the patient will subsequently increase. The training time will be also of 30 minutes

MAINTENANCE CALENDAR (Visits)

RANDOMIZATION visit (V0) (assignment to the maintenance group)

Once completed the intensive treatment of RR, that same day, all patients participating in the trial will be distributed randomly to one of the two groups of RR for maintenance treatment:

-GR1 (TeleRR): will receive an RR of maintenance program with use of support for telemedicine (TeleRR) all of them will be prescribed treatment program at his own home by the doctor, initially very similar to the received in the hospital phase.

Them will be provided the material for the realization of the programme of RR: exercise bike, weights / cufflinks mobile device (PDA/Smartphone) + Pulse Oximeter.

You will indicate them to perform exercises prescribed by your doctor as treatment and that they complete training on the mobile device data. The patient should be sending the data of all the days that are scheduled training exercises once have been completed.

-GR2 (control): receive a recommendation from a standard respiratory rehabilitation program with a minimum monitoring, similar to routine clinical practice.

FOLLOW UP VISITS

In total and after completion of the period of intensive RR, will be planned 3 follow-up visits that may be NO face-to-face or face-to-face and/or ON - LINE:

Visit 1 - tracking: 3 months (± 1 week) after the last visit of randomization (V0).

Visit 2 - follow-up: 9 months (± 2 weeks) after the last visit of randomization (V0).

Visit 3 - follow-up: 12 months (± 2 weeks) after the last visit of randomization (V0), ending the involvement of the patient in the study

NON FACE TO FACE MONITORING

For all visits and patients the participants held a non-contact clinical follow-up through information systems corresponding in each of the participating centres. Information to pick up will be:

If there has been a neglect of the RR maintenance, and if it was so, what have been the causes. If there is a hospital income since the last visit if there is an entry in the emergency room since the last visit If there are visits to unscheduled primary care by exacerbation

FACE TO FACE VISITS

In addition to tracking is not face-to-face, there will be a face-to-face follow-up extraordinary for participating in the trial and that will depend on the group that has been assigned the patient in which the following tests will be carried out:

- Visit 1 -: 3 months (± 1 week) after the last visit of randomization (V0).

Experimental Group GR1:

* Physical examination: weight, height and body mass index.
* Respiratory function tests (spirometry, Lung volumes, transfer to CO, maximum respiratory pressure and blood gas capacity) quality of life health-related questionnaires: CRQ (self-administered version), and SF-36
* Six minutes walking test, assessment of breathlessness to the effort using the Borg scale at the beginning and at the end of six minutes the BODE index calculation test and adverse events or adverse reactions that have been able to present during the period since the previous visit

Visit 2 - follow-up: 9 months (± 2 weeks) after the last visit of randomization (V0):

Experimental Group GR1 :

Physical examination: weight, height and body mass index. Respiratory function tests (spirometry, Lung volumes, transfer to CO, maximum respiratory pressure and blood gas capacity) quality of life health-related questionnaires: CRQ (self-administered version), and SF-36 test of 6 minutes of the March assessment of breathlessness to the effort using the Borg scale at the beginning and at the end of six minutes the BODE index calculation test adverse events or adverse reactions that have been able to present during the period from the previous visit.

Control Group GR2:

• Quality of life health-related questionnaires: CRQ (self-administered version), and SF-36 the 6-minute walking test

- Visit 3 - follow-up: 12 months (± 2 weeks) after the last visit of randomization (V0), where there will be the following

Both Groups GR1 and GR2:

Physical examination: weight, height and body mass index. Respiratory function tests (spirometry, Lung volumes, transfer to CO, maximum respiratory pressure and blood gas capacity) quality of life health-related questionnaires: CRQ (self-administered version), and SF-36 6MWT, assessment of breathlessness to the effort using the Borg scale at the beginning and at the end of six minutes the BODE index calculation test and adverse events or adverse reactions that have been able to present during the period from the previous visit.

ON-LINE FOLLOW UP

Experimental Group GR1

ONLY for patients in the Experimental group, there will be a monitoring On - Line monthly by filling in Telerhabilitacion RR program through the reception of data from the mobile device to the patient

ELIGIBILITY:
Inclusion Criteria:

1. patients with COPD
2. age 8 and 75 (both included)
3. index BODE's 3-7 ( BODE Iindex for Body-mass index, airflow Obstruction, Dyspnea, and Exercise)
4. clinical stability, understood as not having an exacerbation (*) of the COPD and do not require treatment with antibiotics, corticoids systemic and/or hospitalization, at least in the 30 days prior to their inclusion
5. has given his consent
6. capable of using technology
7. the subject is willing and is able to meet all the requirements of the study. * Exacerbation : Exacerbation means worsening of two or more of the following main symptoms for at least 2 consecutive days: dyspnea, volume of sputum; Sputum purulence o worsening of any main symptom along with one of the following symptoms for at least 2 consecutive days: sore throat; Cold ( nasal congestion); Fever without any other cause; Cough; Wheezing

Exclusion Criteria:

1. Osteo-muscular pathology that limit or preclude the exercises
2. Presence of heart disease which limit exercise program
3. patients with bronchiectasis or other several of COPD respiratory disorders
4. comorbidity that prevent respiratory rehabilitation of maintenance program
5. less than 2 years life expectancy
6. any unstable medical or psychiatric process or substance abuse which, in the opinion of the investigator, would affect the ability of the patient to complete the study or impede their participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of an Tele Respiratory Rehabiltation program (TeleRehab) in the maintenance of benefits after an intensive respiratory rehabilitation program evaluated through the 6 m Walking test and health quality questionnaires after 12 months | One Year
  a).Effectiveness of an Tele Respiratory Rehabiltation program in the maintenance of benefits after an intensive respiratory rehabilitation. outcomes:A/ the distancecovered (meters) in the 6m Walking test B/ health quality questionnaires. Specific respiratory questionaire (CRQ); General questionaire (SF 36) after 12 months of maintenance program.C/Changes in the multidimensional scale BODE.
  TeleRR program is clinically effective in the medium and long term by keeping the initial benefits of the intensive RR in aspects such as the capacity of effort (distance in meters), HRQOL and BODE .

SECONDARY OUTCOMES:
Specific objective: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] .Safety of TeleRehab (mortality an serious events due related to the program) | One year
  Safety of TeleRehab defined as directly events related with the program (Injury ,cardiac events, mortality and other events caused during the exercise program),data was recorded in the CRD

OTHER OUTCOMES:
Exploratory objective : To assess the cost effectiveness of the experimental strategy vs the usual approach (Time frame One year) | Two Years
  Exploratory objective : Evaluate the efficiency between the usual approach and experimental strategy (including the TeleRR program) doing an analysis cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: JUAN B GALDIZ ITURRI, PhD, Study Chair — Cruces University Hospital, Biocruces Institute
Locations (1):
- Cruces University Hospital, Biocruces Institute, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galdiz JB, Gomez A, Rodriguez D, Guell R, Cebollero P, Hueto J, Cejudo P, Ortega F, Sayago I, Chic S, Iscar M, Amado C, Rodriguez Trigo G, Cosio BG, Bustamante V, Pijoan JI. Telerehabilitation Programme as a Maintenance Strategy for COPD Patients: A 12-Month Randomized Clinical Trial. Arch Bronconeumol (Engl Ed). 2021 Mar;57(3):195-204. doi: 10.1016/j.arbres.2020.03.034. Epub 2020 May 19. English, Spanish. PMID 32439253